CLINICAL TRIAL: NCT03452956
Title: Cognitive Impairement In Frontotemporal Dementia
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 298201
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Frontotemporal Degeneration; Progressive Supranuclear Palsy; Multiple System Atrophy
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Multiple System Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Cerebral Spinal Fluid (CSF) and blood samples will both be taken and stored for DNA and RNA extraction and analysis and University of Pennsylvania Center for Neurodegenertive Research Center (CNDR).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FTD Cohort: No intervention-observation only
  Interventions: Other: None-Observation Only

INTERVENTIONS:
Other: None-Observation Only — No intervention-this is an observational study

SUMMARY:
This is an observational study that aims to better understand the genetic causes of frontotemporal degeneration (FTD), Multiple Systems Atrophy (MSA), and Progressive Supranuclear Palsy (PSP). It is hoped the information gathered in this study will help lead to better diagnostics and future treatments.

DETAILED DESCRIPTION:
Comparative and longitudinal studies reveal clinical differences between subgroups of patients with frontotemporal dementia (FTD), including Progressive Non-fluent Aphasia (PNFA), Semantic Dementia (SD), patients with a disorder of social comportment and personality (SOC), and non-aphasic patients with executive dysfunction (EXEC). MRI studies of cortical atrophy and fMRI studies show correlated neural defects in FTD subgroups. The investigators will obtain converging evidence from multiple sources to test hypotheses about the neural basis for cognitive functions such as semantic memory, grammatical processing, and social functioning in these FTD subgroups, while improving clinical care for these patients. Recent studies have linked progressive supra nuclear palsy (PSP) and multiple systems atrophy (MSA) to FTD. The investigators will obtain comparable neuropsychological and biomarker data in order to compare these patient groups.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have been diagnosed with FTD, PSP, and MSA

Exclusion Criteria:

* Individuals under 18 years of age
* People with pacemakers or certain metallic implants
* pregnant women

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All individuals with a diagnosis of FTD, PSP, or MSA, previously identified by the PI and sub-investigators through other FTD studies (protocol number 702681) and through the PI's extensive FTD clinical practice at the University of Pennsylvania and at Pennsylvania Hospital's Department of Neurology, will be recruited through letters, brochures, and study flyers.
Sampling Method: Non-Probability Sample
Enrollment: 997 (Actual)
Dates: Start 2003-07-01 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Progression | This is a natural history study - participants are followed from date of enrollment until death, withdrawl, or funding is no longer available, or until 984 months have passed
  Changes over time in MRI and cognitive testing data.

SECONDARY OUTCOMES:
Impaired semantic memory in Semantic Dementia (SD). | This is a natural history study - participants are followed from date of enrollment until death, withdrawl, or funding is no longer available, or until 984 months have passed
  The impact of cortical atrophy on language processing.

OTHER OUTCOMES:
Effortful speech in Progressive Nonfluent Aphasia (PNFA) | This is a natural history study - participants are followed from date of enrollment until death, withdrawl, or funding is no longer available, or until 984 months have passed
  Speech samples related to cortical atrophy seen on MRI and fMRI studies of verb past tense inflection.
Social disinhibition and rule violation in FTD | This is a natural history study - participants are followed from date of enrollment until death, withdrawl, or funding is no longer available, or until 984 months have passed
  Relationship of cognitive testing and MRI data and changes over time.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The University of Pennsylvania is a participant in the National Alzheimer's Coordinating Center 's FTLD-NACC initiative to create a national database of data specific to FTD spectrum diseases.The FTLD NACC initiative will enable research centers focusing on FTD spectrum diseases to gather standardized data on their FTLD patients, all of which will be combined into a single database and made freely available to researchers around the world.
  The FTLD-NACC collects data standardly obtained in this study, including neurocognitive assessments, MRI imaging data, and biomarkers collected through lumbar puncture and blood draw.The FTLD-NACC is designed to facilitate collaborative research and will allow researchers to maximize the use of clinical information and biological material available on frontotemporal degenerative spectrum diseases. Subjects will be able to choose whether or not their research data is shared with the FTD-NACC.
Time Frame: As this is an ongoing, longitudinal study, IPD will be available through the duration of the study.